CLINICAL TRIAL: NCT02247232
Title: Randomized, Double-blind, Placebo-controlled Trial of Z-100 Plus Radiation Therapy in Patients With Locally Advanced Cervical Cancer - A Phase III Trial
Brief Title: Randomized Study of Z-100 Plus Radiation Therapy to Treat Cervical Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Z100-01
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — specific substance maruyama

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Z-100 (Experimental)
  Interventions: Drug: Z-100

INTERVENTIONS:
Drug: Z-100
  Arms: Z-100
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is a phase III, multicenter, double-blind, placebo-controlled, parallel group comparative study to evaluate the efficacy and safety of Z-100 with primary uterine cervical cancer on radiotherapy. The study will use a central randomization with a dynamic allocation using biased coin minimization.

ELIGIBILITY:
Inclusion Criteria:

1. FIGO stage (2008): IIIB, cervical cancer;
2. Pathologically confirmed squamous cell carcinoma of the cervix;
3. Patients with treatment-naive cervical cancer;
4. Patients without enlargement (≥15 mm in the short axis) in the lower abdominal para-aortic lymph node confirmed by CT scanning (Patients need not repeat CT scan at screening if CT data [film or electronic image] within 30 days before informed consent are available and can be provided for central imaging assessment);
5. Patients ≥21, ≤79 years of age at informed consent;
6. Patients for whom it is considered possible to carry out intracavitary radiation in radiotherapy;
7. Eastern Cooperative Oncology Group Performance Status: 0-2;
8. Patients with the following organ functions; (1) WBC ≥3,000/mm3; (2) Platelet count ≥100,000/mm3; (3) Hemoglobin ≥9.5 g/dL (correction by blood transfusion is allowed); (4) Total bilirubin ≤ three (3) times the upper limit of reference value at the clinical testing laboratory; (5) AST, ALT ≤ three (3) times the upper limit of reference value at the clinical testing laboratory; (6) Renal function:

   1. If combination therapy with cisplatin is planned, creatinine clearance: ≥50 mL/min;
   2. If combination therapy with cisplatin is not planned, creatinine ≤ twice (2) the upper limit of reference value at the clinical testing laboratory;
9. Patients who are willing to give informed consents. "

Ages: 21 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 793 (Actual)
Dates: Start 2014-12; Primary Completion 2021-06-29 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5Years

CONTACTS AND LOCATIONS:
Overall Officials: Keiichi Fujiwara, Prof,MD,PhD, Principal Investigator — Saitama Medical University International Medical Center
Locations (7):
- Zeria Invetigative Sites, Tokyo, Japan
- Zeria Investigative Sites, Kuala Lumpur, Malaysia
- Zeria Investigative Sites, Singapore, Singapore
- Zeria Investigative Sites, Seoul, South Korea
- Zeria Investigative Sites, Taipei, Taiwan
- Zeria Investigative Sites, Bangkok, Thailand
- Zeria Investrigative Sites, Hanoi, Vietnam